CLINICAL TRIAL: NCT07380880
Title: Comparison of Proprioceptive Neuromuscular Training and Sensory Re-education in Patients With Diabetic Peripheral Neuropathy
Acronym: PNF-SR in DPN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montiha Azeem (Other)
Responsible Party: Sponsor-Investigator, Montiha Azeem, principal investigator, University of Lahore
Organization: University of Lahore (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOL/IREB/25/15/03/29
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Proprioceptive Neuromuscular Training; Sensory Re-education; Balance; Gait

STUDY DESIGN:
Intervention Model Description: Model Description
Who Masked: Outcomes Assessor
Masking Description: Masking Description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A Sensory Re-Education (Experimental): Participants in this group will receive a structured sensory re-education program for six weeks, with three sessions per week. Each session will include 10 minutes of electrical muscle stimulation (EMS) applied to the lower lumbar region and area of neuropathic discomfort. Sensory re-education will involve stroking the affected skin using brushes and various textured materials, progressing from rough to soft textures over five minutes per session. Balance and gait will be assessed using the Berg Balance Scale (BBS) and Dynamic Gait Index (DGI) at baseline, mid-intervention, and post-intervention.
  Interventions: Behavioral: Sensory Re-Education Program
- group B Proprioceptive Neuromuscular Training (Active Comparator): Participants in this group will undergo a structured proprioceptive neuromuscular training program for six weeks, with three sessions per week. Each session will start with 10 minutes of electrical muscle stimulation (EMS) applied to the lower lumbar region and area of neuropathic discomfort. The main intervention will include balance exercises (bilateral stance, heel raises, single-leg stance with hip flexion, eyes open and closed), strengthening exercises targeting lower limb muscles (quadriceps, hamstrings, lateral thigh), plyometric exercises (single- and double-leg jumps with rotations), and agility drills (figure-eight and directional movements). Each session lasts approximately 30 minutes, and exercises will progress in intensity and complexity based on participant tolerance. Balance and gait outcomes will be measured using the Berg Balance Scale (BBS) and Dynamic Gait Index (DGI) at baseline, mid-intervention, and post-intervention.
  Interventions: Behavioral: Proprioceptive Neuromuscular Training

INTERVENTIONS:
Behavioral: Sensory Re-Education Program — Participants will undergo a six-week sensory re-education program, three sessions per week. Each session includes:
  Electrical Muscle Stimulation (EMS): 10 minutes applied to lower lumbar region and area of neuropathic discomfort (pulse width 100-200 µs, frequency 80-100 Hz, intensity as tolerated).
  Sensory Re-Education: Stroking the affected skin using brushes and textured materials (rough hessian, wool, satin, cotton, fur) for 5 minutes per session, progressing from coarse to soft textures.
  Balance and gait will be assessed using the Berg Balance Scale (BBS) and Dynamic Gait Index (DGI) at baseline, mid-intervention (3 weeks), and post-intervention (6 weeks).
  Arms: group A Sensory Re-Education
Behavioral: Proprioceptive Neuromuscular Training — Participants will receive a structured proprioceptive neuromuscular training program for six weeks, three sessions per week. Each session begins with 10 minutes of electrical muscle stimulation (EMS) applied to the lower lumbar region and area of neuropathic discomfort (pulse width 100-200 µs, frequency 80-100 Hz, intensity as tolerated). The main intervention consists of:
  Balance exercises: bilateral stance, heel raises, single-leg stance with opposite hip flexed, performed with eyes open and closed.
  Strengthening exercises: targeting lower limb muscles including quadriceps, hamstrings, and lateral thigh using squats and resistance exercises.
  Plyometric exercises: single- and double-leg jumps with 90° and 180° rotations to enhance coordination.
  Agility drills: figure-eight running and directional movements (forward, backward, lateral) along straight and spiral paths.
  Each session lasts approximately 30 minutes, with progressive intensity and complexity based on individual toleran
  Arms: group B Proprioceptive Neuromuscular Training

SUMMARY:
Diabetic peripheral neuropathy (DPN) is a common complication of diabetes mellitus and is associated with sensory loss, impaired proprioception, balance deficits, and altered gait patterns, which significantly increase the risk of falls and functional dependence. Rehabilitation strategies targeting sensory and proprioceptive impairments are essential to improve postural control and mobility in this population.

This randomized controlled trial aims to compare the effects of proprioceptive neuromuscular training and sensory re-education on balance and gait performance in patients with diabetic peripheral neuropathy. Participants diagnosed with DPN will be randomly allocated into two groups. Group A will receive sensory re-education, while Group B will undergo a structured proprioceptive training program. Both groups will also receive baseline conventional treatment.

Balance and gait outcomes will be assessed using the Berg Balance Scale and the Dynamic Gait Index at baseline, mid-intervention, and post-intervention. The findings of this study may help determine the more effective rehabilitation approach for improving balance and gait in individuals with diabetic peripheral neuropathy, thereby reducing fall risk and enhancing functional independence.

DETAILED DESCRIPTION:
Diabetic peripheral neuropathy is a progressive complication of diabetes characterized by sensory impairment, proprioceptive deficits, and neuromuscular dysfunction. These impairments adversely affect balance control and gait stability, increasing the likelihood of falls, injuries, and reduced quality of life. Despite the widespread use of rehabilitation interventions, there is limited comparative evidence regarding the effectiveness of sensory re-education versus proprioceptive neuromuscular training in improving functional outcomes among individuals with DPN.

This randomized controlled trial will be conducted at the University Institute of Physical Therapy, Lahore, following approval from the Institute Research Ethics Board. Eligible participants with confirmed diabetic peripheral neuropathy will be recruited through referrals from endocrinologists and diabetologists. After obtaining informed consent, participants will be randomly assigned to either the sensory re-education group or the proprioceptive training group using a lottery method. The study will follow a single-blinded design, with outcome assessors blinded to group allocation.

Both groups will undergo a six-week intervention program consisting of three supervised sessions per week. Balance and gait performance will be evaluated at baseline, at the third week, and at the completion of the intervention using standardized outcome measures. Data analysis will focus on comparing within-group and between-group changes over time.

The results of this study are expected to provide evidence-based guidance for physical therapists in selecting effective rehabilitation strategies to improve balance and gait in patients with diabetic peripheral neuropathy, ultimately aiming to reduce fall risk and enhance functional mobility.

ELIGIBILITY:
Inclusion Criteria:

Both males and females Diagnosed with Diabetes Mellitus (Type 1 or Type 2) Aged between 40-75 years Presence of diabetic peripheral neuropathy (as confirmed by Michigan Neuropathy Assessment Tool or Toronto Clinical Rating Scale) HbA1c level > 7% consistently over the last 6 months

Exclusion Criteria:

Unable to ambulate independently or with assistance Any history of neurological disorders Any history of musculoskeletal disordersin the past 6 months Renal and liver failure History of Ischemic heart disease History of dizziness or balance-impairing conditions

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Balance Performance Assessed by the Berg Balance Scale | Baseline, 3 weeks, and 6 weeks after the start of intervention
  The primary outcome is the change in balance performance in patients with diabetic peripheral neuropathy. Balance will be measured using the Berg Balance Scale (BBS), a validated tool consisting of 14 tasks evaluating both static and dynamic balance, scored from 0 (lowest function) to 4 (best performance), with a total maximum score of 56. Higher scores indicate better balance and mobility. Assessments will be conducted at baseline, at 3 weeks, and at 6 weeks post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Nimra Zaheer, MSPTN, Principal Investigator — The University of Lahore, Lahore
Locations (1):
- Shadman Medical Center, Lahore, Punjab Province, Pakistan